CLINICAL TRIAL: NCT05528900
Title: Pathways of Children With Food Protein Induced Enterocolitis Syndrome in Its Acute Form : a Multicentre Prospective Study - National FPIES Observatory
Brief Title: A Multicentre French Prospective Study of Children With Food Protein Induced Enterocolitis Syndrome in Its Acute Form
Acronym: SEIPA-FPIES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Lenval (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-HPNCL-03
Record Dates: First submitted 2022-07-29; First posted 2022-09-06 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-03

CONDITIONS: Food Protein Induced Enterocolitis Syndrome (FPIES)
Keywords: Non IgE mediated food allergy; FPIES,; children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FPEIS children (Experimental)
  Interventions: Diagnostic Test: allergy test

INTERVENTIONS:
Diagnostic Test: allergy test — allergy test are oral food challenge , prick test and IgE blood rate

SUMMARY:
Food protein induced enterocolitis syndrome (FPIES), is a non-IgE mediated food allergy (FA) which seems to expand, and occurring in infancy. This disease is usually unknown by clinicians. In 2017, an international workgroup of American Academy of Allergy, Asthma and Immunology published clinical criteria to specify the diagnosis. However, there is a lack of information in literature for describe the evolution and atypical phenotypes. In addition, no prospective French series has been published to date. The aim of the study is to collect clinical features and allergy testing of children who have acute form of FPIES at diagnosis and during evolution during three years

DETAILED DESCRIPTION:
Food protein induced enterocolitis syndrome (FPIES), is a non-IgE mediated food allergy (FA) which seems to expand, and occurring in infancy. Prevalence of FPIES is unknown. In 2011, Katz published cumulative incidence of cow 'milk FPIES of 3 per 1000 new-borns, from prospective birth cohort in Israel.

The offending food depend on the country, probably in relation to eating habits.

Cow's milk (CM) is most commonly incriminated and can lead to a chronic digestive disease or in its acute form with potentially life-threatening vomiting/diarrhoea/dehydration, confusing with anaphylaxis. Rice and oat in US, or fish and egg in France are the solid food most often implicated.

This disease is usually unknown by clinicians. Its diagnostic is based on clinical history, and differential diagnosis elimination.

In 2017, an international workgroup of American Academy of Allergy, Asthma and Immunology published clinical criteria to specify the diagnosis and management. According to this last definition (JACI 2017), patient have to meet the major criterion and at least 3 minor criteria. Major criterion is vomiting in the 1- to 4-h period after ingestion of the suspect food and absence of classic IgE-mediated allergic skin or respiratory symptoms. Minor criteria are :

1. A second (or more) episode of repetitive vomiting after eating the same suspect food,
2. Repetitive vomiting episode 1-4 h after eating a different food
3. Extreme lethargy with any suspected reaction
4. Marked pallor with any suspected reaction
5. Need for emergency department visit with any suspected reaction
6. Need for intravenous fluid support with any suspected reaction
7. Diarrhea in 24 h (usually 5-10 h)
8. Hypotension
9. Hypothermia Skin prick test et IgE antibody are negative except atypical FPIES. Acute management begins with clinical evaluation, then administer normal saline bolus quickly. Parenteral ondansetron can be used to stop vomiting. Nutritional management implicate elimination of the offending foods. Only the oral food challenge in hospital can be done to determine resolution of FPIES after a long time of no symptom.

The age of tolerance, depend of the food. The average age of acquiring tolerance for cow's milk changes in the literature, around 8-10 months in Korea, around 1 year in Israel, around 5 years in the United States. There is no data in France on the recovery age of CM-FPIES.

However, there is a lack of information in literature for describe the evolution and atypical phenotypes. In addition, no prospective French series has been published to date.

Our work is a national prospective study, which will collect news cases of acute FPIES diagnosis in sixteen French centres.

Main objective: To determine the rate of acquisition of tolerance by food at 1 year, 2 years, 3 years post inclusion.

Secondary objectives:

* Description of a population of children with newly diagnosed FPIES. 2. Describe the rate of patients with FPIES progressing to IgE sensitization whatever the food at 1 year, 2 years, 3 years post inclusion.

  3. Determine per food the rate of FPIES patients evolving towards IgE sensitization at 1 year, 2 years, 3 years post inclusion.

  4. Describe the rate of patients with FPIES progressing to clinical symptoms of IgE-mediated allergy, whatever the food, at 1 year, 2 years, 3 years post inclusion.

  5. Determine, by food, the rate of FPIES evolving towards clinical symptoms of IgE-mediated allergy at 1 year, 2 years, 3 years post inclusion.

  6. Describe the rate of patients with multiple FPIES at each time point of the study.

  7. Describe at each time the rates of patients with personal atopic comorbidities.

The inclusion period will last three years, and the follow up of each patient will last three years.

Allergologist will see the patient at inclusion visit, then one time a year. If the patient does not acquire tolerance, an oral food challenge (OFC) in hospital will lead to answer.

The aim of our work will help allergologist to manage FPIES children, with French specificities in offending food, and tolerance.

ELIGIBILITY:
Inclusion Criteria:

* age from 0 to 17 years old,
* seen in allergologist visit for acute FPIES, due to history of suggestive clinical symptoms, confirmed by the criteria published in 2017 in the JACI (Nowak-Wegrzyn et al, JACI 2017), or by an oral food challenge for diagnosis in the absence of the requested clinical criteria,
* affiliated to social security (public healthcare system)
* signed consent of one of the parents or the holder of parental authority

Exclusion Criteria:

* Associated pathology that may contraindicate OFC at the discretion of the investigating physician. In particular justifying permanent treatment with a beta-blocker or an angiotensin-converting enzyme inhibitor.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
tolerance acquisition | through study completion, an average of 6 years
  The acquisition of tolerance will be defined by negative OFC or accidental intake of the food at home tolerated according to parents discussion

SECONDARY OUTCOMES:
population description | through study completion, an average of 6 years
  The description of the population included will be made according to the clinical, the demographic data, the allergy tests, the history of the disease
IgE sensitization | at 1 year, 2 years, 3 years post inclusion
  IgE sensitization is defined by the positivity of an immediate-read skin test (wheal of the prick test greater than half of the positive histamine control) and/or the presence of specific IgE antibody on a blood sample (≥0.35 kU/L).
food sensitization | at 1 year, 2 years, 3 years post inclusion
  food sensitization is defined by the positivity of an immediate-read skin test (wheal of the prick test greater than half of the positive histamine control)
IgE-mediated allergy | at 1 year, 2 years, 3 years post inclusion
  IgE-mediated allergy is defined by the demonstration of clinical symptoms related to the presence of these specific IgEs.
IgE-dependent allergy | at 1 year, 2 years, 3 years post inclusion
  IgE-dependent allergy will be defined by the appearance of symptoms a few minutes to 2 hours after ingestion of the food, with skin signs (urticaria, angioedema) and/or respiratory symptoms (dyspnea, laryngospasm, cough, bronchospasm ); digestive and neurological signs being potentially common with the diagnosis of FPIES
multiple FPIES | at 1 year, 2 years, 3 years post inclusion
  A multiple FPIES will be defined by the presence of clinical symptoms of FPIES for at least two different foods
Atopic comorbidities | at 1 year, 2 years, 3 years post inclusion
  Atopic comorbidities will be defined by asthma, allergic rhinitis, atopic dermatitis, and eosinophilic esophagitis

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - Chu Angers, Angers
  - Chi Robert Ballanger, Aulnay-sous-Bois
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - Hopital Civils de Colmar, Colmar
  - Chu Grenoble, Grenoble
  - Ch Haguenau, Haguenau
  - Chr Lille Hopital Jeanne de Flandre, Lille
  - Hopital Saint Vincent de Paul Ghicl, Lille
  - Hopital Civil de Lyon, Lyon
  - Chu Montpellier, Montpellier
  - Chu Nancy, Nancy
  - Cabinet Berlioz, Nice
  - Hôpitaux Pédiatriques de Nice CHU-Lenval, Nice
  - Aphp Armand Trousseau, Paris
  - Hopital Ambroise Pare Aphp, Paris
  - Hopital Necker Enfants Malades Aphp, Paris
  - Hopital Robert Debre Aphp, Paris
  - Chu Rouen, Rouen
  - Cabinet Chabbert, Toulouse